CLINICAL TRIAL: NCT05450172
Title: Impact of Postoperative Transitional Pain on Recovery After Thoracic Surgery
Acronym: TRANSAT
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC22_0203
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Recovery
Keywords: Postoperative transitional pain; postoperative pain trajectory; postoperative neuropathic pain; thoracic surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consecutive patients scheduled for thoracic surgery
  Interventions: Other: QoR-15 questionnaire

INTERVENTIONS:
Other: QoR-15 questionnaire — The QoR-15 is a 15-item questionnaire on postoperative quality of recovery. The DN4 is a 10-item questionnaire on neuropathic pain. Both questionnaires will be given to the patients preoperatively, on postoperative days 2 and 3, and 1, 3 and 6 months after surgery.
  Other Names: DN4 questionnaire

SUMMARY:
Postoperative transitional pain corresponds to the pain occuring between acute postoperative pain and chronic postsurgical pain (defined as pain persisting for at least 3 months after surgery). We hypothesized that both trajectory and neuropathic component of transitional pain may influence the quality of recovery after thoracic surgery. To test this, we designed an observational study to identify risk factors for incomplete recovery assessed through the QoR-15 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* patients scheduled for thoracic surgery (thoracotomy or video-assisted thoracic surgery or surgery for thoracic outlet syndrome)
* patients who do not object to the study

Exclusion Criteria:

* patients non francophone
* emergency surgery or revision surgery
* patients already included in the study during the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for thoracic surgery (thoracotomy or video-assisted thoracic surgery or surgery for thoracic outlet syndrome).
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Impact of pain trajectory and neuropathic component of pain on quality of recovery. | 3 months after surgery.
  An incomplete recovery will be defined as a postoperative QoR-15 score of at least 8 points lower than the preoperative QoR-15 value. The association between both trajectory and neuropathic component of postoperative transitional pain and incomplete recovery will be evaluated.

SECONDARY OUTCOMES:
Description of trajectory and neuropathic component of postoperative transitional pain. | Between postoperative day 2 and 3 months after surgery.
  To describe the trajectory and neuropathic component of postoperative transitional pain according to QoR-15 and DN4 successive values.
Impact of the type of surgery on quality of recovery. | 3 months after surgery.
  To assess the impact of thoracotomy or video-assisted thoracic on quality of recovery.
Impact of pain trajectory, neuropathic component of pain and type of surgery on chronic postsurgical pain prevalence. | 3 and 6 months after surgery.
  To assess the impact pain trajectory, neuropathic component of pain and type of surgery on chronic postsurgical pain prevalence.
Predictive accuracy of neuropathic pain trajectory on incomplete recovery and chronic postsurgical pain prevalence. | 3 and 6 months after surgery.
  To assess the predictive accuracy of neuropathic pain trajectory on incomplete recovery and chronic postsurgical pain prevalence.
Correlation between neuropathic componente of chronic postsurgical pain and quality of recovery. | 3 and 6 months after surgery.
  To assess the correlation between neuropathic componente of chronic postsurgical pain and quality of recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided